CLINICAL TRIAL: NCT01102569
Title: Molecular Genetics and Epidemiology of Pancreatic Cancer in Ashkenazi Jewish Patients
Brief Title: Pancreatic Cancer Genetics
Status: Recruiting | Type: Observational
Sponsor: Columbia University (Other)
Responsible Party: Sponsor
Other Study IDs: AAAC6344
Record Dates: First submitted 2010-04-12; First posted 2010-04-13 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-04

CONDITIONS: Pancreatic Cancer
Keywords: Hereditary pancreatic cancer; Breast and Ovarian Cancer Syndrome; BRCA1/2; Ashkenazi Jewish patients
MeSH Terms: conditions — Pancreatic Neoplasms; Pancreatic carcinoma, familial

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Peripheral Blood Specimens: Three tubes of blood will be collected from each study participant. A portion of the blood will be utilized to extract white blood cells that will be immortalized by Epstein-Barr virus (EBV) infection.
  * Archived Fixed Tissue Samples: Tissue blocks from surgery performed at Columbia University Medical Center or elsewhere, will be requested after obtaining consent for study participation.
  * Fresh Tissue Collection: At the time of surgery for tumor resection, tumor and adjacent normal tissue will be requested from the Pathology Department. At the time of endoscopy, aspirated fluid or biopsied tissue will be requested. No additional tissue will be resected beyond that required for surgical or endoscopic management.
  * Genetic Testing: Genetic testing will be performed in a New York State certified research laboratory . Test results from research laboratories will not be disclosed to patients.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Pancreatic cancer and Ashkenazi decent: Patients with pancreatic cancer will be asked to join the study if they identify themselves as being of Ashkenazi descent, as well as patients at a high-risk of pancreas cancer based on family history, and will be followed from the time of diagnosis.

SUMMARY:
The aim of this study is to determine the frequency of the three most common BReast CAncer gene 1 (BRCA1) and BReast CAncer gene 2 (BRCA2) genetic mutations that are commonly found in Ashkenazi Jewish patients with pancreatic cancer. Testing for BRCA1 and BRCA2 mutations in relatives of hereditary pancreatic cancer patients may have a significant impact; allowing for early screening, treatment, and resection of pre-malignant tissue or malignant lesions.

DETAILED DESCRIPTION:
Pancreatic cancer is the fourth leading cause of death from malignancy in the United States. Up to 15% of pancreatic cancers have a hereditary component. Several gene mutations and cancer syndromes have been identified that are frequently found in greater frequency in individuals with pancreatic cancer, including the breast ovary cancer syndrome (BRCA1/BRCA2 mutations). No studies adequately describe the epidemiology of inherited pancreatic cancer and genetic risk factors that may modify the penetrance of BRCA1/BRCA2 mutations. The primary aim of this study is to determine the frequency of BRCA1 (185delAG,5382insC) and BRCA2 (6174delT) mutations in Ashkenazi Jewish pancreatic cancer patients. Secondary endpoints will include determining the individual frequency of these mutations and other disease-modifying mutations, death from any cause, disease-free survival, and stage of disease at time of presentation, differences in tissue pathology, risk factors, treatment decisions and development of metachronous malignancies.

The investigator plans to study about 100 patients, which will enable the true frequency of the mutation to be estimated. Although the impact of BRCA1/BRCA2 mutations will be initially studied in the Ashkenazi population, these data will be widely applicable to other pancreatic cancer patients carrying BRCA1/BRCA2 mutations. Testing for BRCA1 and BRCA2 mutations in relatives of hereditary pancreatic cancer patients may allow early screening, treatment, and resection of pre-malignant tissue or malignant lesions.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with pancreatic cancer.
* Patients are of Ashkenazi Jewish descent.
* Patients have been Columbia Pancreatic Cancer Prevention Program Registry and Tissue Bank for High-Risk Individuals (IRB-AAAA6154).

Exclusion Criteria:

* Inability to provide informed consent.
* Under the age of 18 years old.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study subjects will be pancreatic cancer patients at CUMC who are of Ashkenazi Jewish descent.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2008-01; Primary Completion 2026-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of Three BRCA1/2 Mutations in Ashkenazi Jewish Patients | 1 year
  The primary aim of this study is to determine the combined frequency of BRCA1 (185delAG, 5382insC) and BRCA2(6174delT) mutations in Ashkenazi Jewish pancreatic cancer patients.

SECONDARY OUTCOMES:
Individual Frequency of Three Mutations | 1 year
  Individual frequency of these mutations three mutations BRCA1 (185delAG, 5382insC) and BRCA2 (6174delT) mutations.
Frequency of disease modifying mutations | 1 year
  Determine the frequency of disease modifying mutations such as MSH2 A636P, APC I1307K, P53, R72P, CHEK2 S428F, RAD51 G135C and MTHFR V222A.

CONTACTS AND LOCATIONS:
Overall Officials: Fay Kastrinos, MD, Principal Investigator — Columbia University
Locations (1):
- Columbia University Medical Center, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No